CLINICAL TRIAL: NCT02852252
Title: Solid Tumor Cancer Surgery With or Without Intraoperative Imaging: A Registry Optional Sub-Study I: ICG Optional Sub-Study II: OTL38
Brief Title: Solid Tumor Cancer Surgery With or Without Intraoperative Imaging: A Registry
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 822933
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Bladder Cancer; Gastric Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Stomach Neoplasms | interventions — Pafolacianine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: OTL38 — Patients will be given imaging agent 2-3 hours before surgery to assist in imaging.
Drug: ICG — Patients will be given imaging agent 24 hours before surgery to assist in imaging.

SUMMARY:
The study objective is to collect prospective data on cancer patients who undergo surgery and intraoperative imaging. The registry will include (but not limited to) cancer type, stage, intraoperative challenges to the surgeon, usage and results of intraoperative imaging, and recurrence surveillance.

DETAILED DESCRIPTION:
Our objective is to collect prospective data on cancer subjects who undergo surgery and intraoperative imaging. The registry will include (but not limited to) cancer type, stage, intraoperative challenges to the surgeon, usage and results of intraoperative imaging, and recurrence surveillance.

In this protocol, subjects that receive intraoperative imaging will provide us the opportunity to record what tissues fluoresce in the operating room, and then to identify if these lesions are cancer when the histopathology is performed. Also, we will monitor any side effects or potential toxicities that may occur. This data can then be used to predict if a subject is more likely to develop a local recurrence due to missed cancer cells, metastatic lymph nodes or synchronous lesions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >/= 18 years of age.
* Patients presenting with esophagogastric or bladder cancer.
* Good operative candidate as determined by the treating physician and/or multidisciplinary team.
* Subject capable of giving informed consent and participating in the process of consent.

Exclusion Criteria:

* Pregnant women as determined by urinary or serum beta hCG within 72 hours of surgery.
* Vulnerable patient population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a high clinical suspicion of cancer, scheduled to undergo surgery.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Tissue to Background Ratio | 2 years
  Enhance ability to detect malignant tissues in situ and ex vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States